CLINICAL TRIAL: NCT01239823
Title: Platform Exercise Training for Women at Risk for Knee Osteoarthritis
Brief Title: Platform Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Neil A. Segal, MD, The University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N2009120009
Record Dates: First submitted 2010-11-02; First posted 2010-11-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; whole body vibration; mobility; rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Exercise; Vibration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Body Vibration Training (Experimental): The subjects will participate in a 12-week whole body vibration exercise program with 2 sessions (1/2 hour) per week.
  Interventions: Other: Whole Body Vibration Training
- Exercise without vibration (Experimental): The subjects will participate in a 12-week exercise program with 2 sessions (1/2 hour) per week.
  Interventions: Other: Exercise without vibration

INTERVENTIONS:
Other: Whole Body Vibration Training — The subjects will participate in a 12-week exercise program with two sessions (1/2 hour) per week.
  Arms: Whole Body Vibration Training
Other: Exercise without vibration — Participants will complete the same exercises without vibration twice a week for 12 weeks (1/2 hour sessions).
  Arms: Exercise without vibration

SUMMARY:
The purpose of this randomized, controlled trial is to determine whether a vibration platform exercise program will be more effective than a standard platform exercise program in improving quadriceps strength in women age 45-60 who have risk factors for knee osteoarthritis. Each platform exercise program will be conducted 2 times a week for 12 weeks. The sessions will consist of a series of exercises on a Wave Pro-elite vibration platform (with 1-3 minute rests between sets) and stretches with the platform vibration either turned on (intervention group) or off (control group.) Quadriceps strength (primary outcome), leg press power, and vibration sense will be assessed at baseline and 12 weeks, and changed scores will be compared between groups.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common disabling disease in older adults,(1) affecting over 25 million Americans, resulting in significantly impaired function and mobility(2) and a societal economic burden.(3) The knee is the weight-bearing joint most commonly affected,(10) and the prevalence of symptomatic knee OA is between 9% and 21% among those 65 years and older.(2, 11, 21) Loss of knee range of motion can lead to significant difficulty in bathing, lower body dressing, stair mobility, and walking.

Impaired mobility due to knee OA will have an increasingly significant societal impact, with 67 million adults projected to have arthritis by 2030, and 25 million with arthritis-attributable activity limitations.(22) Women are at greater risk for knee OA compared with men. Knee OA leads to chronic disability,(23-25) functional limitations,(26) and dependence.(27) Patients with knee OA frequently are limited in their activities by joint stiffness or buckling, decreased range of motion, muscle weakness, poor balance, impaired proprioception, reduced vibration sense, and/or pain. Currently, there are limited options available for patients for improving the outcome of knee OA once they have it. At this time, patients may use analgesics for pain with total knee replacement as the last option. However, we recently found that greater quadriceps strength protected against the development of incident symptomatic knee OA and progression of knee OA in women.(19-20) Thus, strengthening the quadriceps muscle may prevent worsening of the knee joint. Though before studying whether strengthening is effective in reducing risk for knee OA, it is necessary to first determine an effective and tolerated means of exercise.

Vibration platform exercise may provide the benefits of strength training without adding potentially harmful loads to the knee joint. In one study of nursing home residents with limited functional capacity, balance and mobility improved over a 6-week whole body vibration exercise program. (12) In another study that compared whole body vibration (WBV) to resistance training in older women, greater improvement in knee extensor strength and speed of movement was found with WBV exercise.(13) Additionally, after a 2-month exercise program with older adults between the ages of 59 to 86, walking speed, step length, and the maximum standing time on one leg significantly improved with WBV exercise.(14) WBV exercise was safe and well tolerated in the elderly.(14, 15, 16) There have also been indications that WBV may improve flexibility. While a study testing range of motion (ROM) found that both the WBV and the control groups had significant increases in hamstring flexibility, only the WBV group showed a significantly larger increase (30%) in ROM than did the control group (14%).(17) There have also been indications WBV may improve proprioception (joint position sense) in women with knee osteoarthritis. One study which compared control versus exercise on a vibration platform and a balance board vibration platform found improvements in muscle strength and proprioception, respectively.(18) Thus, these studies suggest a beneficial effect of WBV exercise in addition to muscle strengthening, balance, and walking exercises in improving the walking ability in the elderly.

Exercises conducted on a vibrating platform will induce a muscle reflex, increasing muscle fiber activation at a higher level compared to performing the exercises on a non-vibrating platform. We have selected the frequency and duration of this program based on 1) frequency used in previous studies and recommended by the manufacturer and 2) duration of 12 weeks based on previous data which found the most gain in knee extensor strength and speed of the movement occurred at week 12 of a 24-week program. (13)

Vibration exercise may be a better option than strength training alone, if the exercises can be completed in less time and with similar strength gains as resistance training, but without the additional loads contributing to the stress on patients' joints.

ELIGIBILITY:
Inclusion Criteria:

* age 45-60
* female
* history of knee injury or surgery (except replacement surgery) or body mass index (BMI) greater than or equal to 25.

Exclusion Criteria:

* diagnosis of knee osteoarthritis
* inflammatory arthritis such as rheumatoid or psoriatic arthritis
* knee replacement
* metallic implant or stent placement surgery or any implanted devices
* surgery or lower limb injury in the last 6 months that affects walking ability
* lower limb amputation (other than single ray)
* unable to walk without an assistive device
* wounds that contraindicate weight-bearing exercise
* acute infection or inflammation that contraindicates exercise
* acute disk related problems (new lower back pain in the last 3 months or severe enough to affect walking)
* osteonecrosis
* currently pregnant or planning to become pregnant
* kidney, bladder or gallstones that have not been passed
* retinal detachment
* ever experienced deep vein thrombosis
* type 1 diabetes mellitus (insulin dependent)
* history of myocardial infarction or stroke in the last year
* medical conditions that affect walking ability or ability to take part in the study or exercise such as; Alzheimer's disease, multiple sclerosis, Parkinson's disease, severe cardiovascular disease, congestive heart failure, severe emphysema, severe asthma, severe dysrhythmias or pacemaker
* Any type of implanted pump (e.g. Morphine, baclofen) or catheter (e.g. In kidney, brain or spine)
* neuropathy (by Semmes-Weinstein Monofilament)
* uncontrolled epilepsy
* active cancer (< 5 years since remission) or other illness expected to be terminal within 1 year
* concurrent participation in another research study
* Inability to follow protocol (e.g. lack of ability to attend visits or understand instructions)
* frequent knee pain on most of the last 30 days

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Isokinetic quadriceps strength | Change from baseline to 12 weeks

SECONDARY OUTCOMES:
Vibration Perception Threshold | Change from baseline to 12 weeks
Leg press muscle power | Change from baseline to 12 weeks
Timed Stair Climb | Change from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] The American Geriatrics Society. Research and Geriatric Medicine Position Statement. http://www.americangeriatrics.org/products/positionpapers/research.shtml ed. New York: AGS Public Policy Committee; 1999.
- [Background] Nevitt MC, Lane N. Body weight and osteoarthritis. Am J Med. 1999 Dec;107(6):632-3. doi: 10.1016/s0002-9343(99)00297-1. No abstract available. PMID 10625033
- [Background] March LM, Bachmeier CJ. Economics of osteoarthritis: a global perspective. Baillieres Clin Rheumatol. 1997 Nov;11(4):817-34. doi: 10.1016/s0950-3579(97)80011-8. PMID 9429738
- [Background] Guccione AA. Arthritis and the process of disablement. Phys Ther. 1994 May;74(5):408-14. doi: 10.1093/ptj/74.5.408. PMID 8171102
- [Background] Kramer JS, Yelin EH, Epstein WV. Social and economic impacts of four musculoskeletal conditions. A study using national community-based data. Arthritis Rheum. 1983 Jul;26(7):901-7. doi: 10.1002/art.1780260712. PMID 6223644
- [Background] Hurley MV. The role of muscle weakness in the pathogenesis of osteoarthritis. Rheum Dis Clin North Am. 1999 May;25(2):283-98, vi. doi: 10.1016/s0889-857x(05)70068-5. PMID 10356418
- [Background] McGibbon CA, Krebs DE, Scarborough DM. Rehabilitation effects on compensatory gait mechanics in people with arthritis and strength impairment. Arthritis Rheum. 2003 Apr 15;49(2):248-54. doi: 10.1002/art.11005. No abstract available. PMID 12687518
- [Background] Felson DT. Epidemiology of hip and knee osteoarthritis. Epidemiol Rev. 1988;10:1-28. doi: 10.1093/oxfordjournals.epirev.a036019. PMID 3066625
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of self-reported arthritis or chronic joint symptoms among adults--United States, 2001. MMWR Morb Mortal Wkly Rep. 2002 Oct 25;51(42):948-50. PMID 12437034
- [Background] Davis MA. Epidemiology of osteoarthritis. Clin Geriatr Med. 1988 May;4(2):241-55. PMID 3288318
- [Background] Andersen RE, Crespo CJ, Ling SM, Bathon JM, Bartlett SJ. Prevalence of significant knee pain among older Americans: results from the Third National Health and Nutrition Examination Survey. J Am Geriatr Soc. 1999 Dec;47(12):1435-8. doi: 10.1111/j.1532-5415.1999.tb01563.x. PMID 10591238
- [Background] Bautmans I, Van Hees E, Lemper JC, Mets T. The feasibility of Whole Body Vibration in institutionalised elderly persons and its influence on muscle performance, balance and mobility: a randomised controlled trial [ISRCTN62535013]. BMC Geriatr. 2005 Dec 22;5:17. doi: 10.1186/1471-2318-5-17. PMID 16372905
- [Background] Roelants M, Delecluse C, Verschueren SM. Whole-body-vibration training increases knee-extension strength and speed of movement in older women. J Am Geriatr Soc. 2004 Jun;52(6):901-8. doi: 10.1111/j.1532-5415.2004.52256.x. PMID 15161453
- [Background] Kawanabe K, Kawashima A, Sashimoto I, Takeda T, Sato Y, Iwamoto J. Effect of whole-body vibration exercise and muscle strengthening, balance, and walking exercises on walking ability in the elderly. Keio J Med. 2007 Mar;56(1):28-33. doi: 10.2302/kjm.56.28. PMID 17392595
- [Background] Bruyere O, Wuidart MA, Di Palma E, Gourlay M, Ethgen O, Richy F, Reginster JY. Controlled whole body vibration to decrease fall risk and improve health-related quality of life of nursing home residents. Arch Phys Med Rehabil. 2005 Feb;86(2):303-7. doi: 10.1016/j.apmr.2004.05.019. PMID 15706558
- [Background] Bogaerts A, Verschueren S, Delecluse C, Claessens AL, Boonen S. Effects of whole body vibration training on postural control in older individuals: a 1 year randomized controlled trial. Gait Posture. 2007 Jul;26(2):309-16. doi: 10.1016/j.gaitpost.2006.09.078. Epub 2006 Oct 30. PMID 17074485
- [Background] van den Tillaar R. Will whole-body vibration training help increase the range of motion of the hamstrings? J Strength Cond Res. 2006 Feb;20(1):192-6. doi: 10.1519/R-17064.1. PMID 16503680
- [Background] Trans T, Aaboe J, Henriksen M, Christensen R, Bliddal H, Lund H. Effect of whole body vibration exercise on muscle strength and proprioception in females with knee osteoarthritis. Knee. 2009 Aug;16(4):256-61. doi: 10.1016/j.knee.2008.11.014. Epub 2009 Jan 15. PMID 19147365
- [Background] Segal NA, Glass NA, Torner J, Yang M, Felson DT, Sharma L, Nevitt M, Lewis CE. Quadriceps weakness predicts risk for knee joint space narrowing in women in the MOST cohort. Osteoarthritis Cartilage. 2010 Jun;18(6):769-75. doi: 10.1016/j.joca.2010.02.002. Epub 2010 Feb 11. PMID 20188686
- [Background] Segal NA, Torner JC, Felson D, Niu J, Sharma L, Lewis CE, Nevitt M. Effect of thigh strength on incident radiographic and symptomatic knee osteoarthritis in a longitudinal cohort. Arthritis Rheum. 2009 Sep 15;61(9):1210-7. doi: 10.1002/art.24541. PMID 19714608
- [Background] Felson DT. The epidemiology of knee osteoarthritis: results from the Framingham Osteoarthritis Study. Semin Arthritis Rheum. 1990 Dec;20(3 Suppl 1):42-50. doi: 10.1016/0049-0172(90)90046-i. PMID 2287948
- [Background] Hootman JM, Helmick CG. Projections of US prevalence of arthritis and associated activity limitations. Arthritis Rheum. 2006 Jan;54(1):226-9. doi: 10.1002/art.21562. PMID 16385518
- [Background] Fried LP, Bandeen-Roche K, Chaves PH, Johnson BA. Preclinical mobility disability predicts incident mobility disability in older women. J Gerontol A Biol Sci Med Sci. 2000 Jan;55(1):M43-52. doi: 10.1093/gerona/55.1.m43. PMID 10719772
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Ling SM, Fried LP, Garrett ES, Fan MY, Rantanen T, Bathon JM. Knee osteoarthritis compromises early mobility function: The Women's Health and Aging Study II. J Rheumatol. 2003 Jan;30(1):114-20. PMID 12508399
- [Background] Davis MA, Ettinger WH, Neuhaus JM, Mallon KP. Knee osteoarthritis and physical functioning: evidence from the NHANES I Epidemiologic Followup Study. J Rheumatol. 1991 Apr;18(4):591-8. PMID 2066950
- [Background] Guccione AA, Felson DT, Anderson JJ. Defining arthritis and measuring functional status in elders: methodological issues in the study of disease and physical disability. Am J Public Health. 1990 Aug;80(8):945-9. doi: 10.2105/ajph.80.8.945. PMID 2368855